CLINICAL TRIAL: NCT03426124
Title: Retrospective and Prospective International EkoSonic® Registry of the Treatment and Clinical OUTcomes of Patients With Pulmonary Embolism
Brief Title: An International Pulmonary Embolism Registry Using EKOS
Acronym: KNOCOUT PE
Status: Completed | Type: Observational
Sponsor: Boston Scientific Corporation (Industry)
Collaborators: BTG International Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: BTG-001653-01
Record Dates: First submitted 2018-01-29; First posted 2018-02-08 (Actual); Results first posted 2023-02-22 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2022-05

CONDITIONS: Pulmonary Embolism and Thrombosis
Keywords: venous thromboembolism
MeSH Terms: conditions — Pulmonary Embolism; Thrombosis; Venous Thromboembolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- Retrospective: Individuals with intermediate-high or high risk pulmonary embolism who were consecutively treated with the Ekosonic Endovascular System (EKOS) and thrombolytic drug between January 2014 and one year prior to site activation.
  Interventions: Device: EkoSonic Endovascular System with thrombolytic
- Prospective: Individuals who are experiencing intermediate-high or high risk pulmonary embolism where the treating investigator has selected the EKOS device and thrombolytic drug. The duration of ultrasound and volume of thrombolytic drug are selected per physician discretion.
  Interventions: Device: EkoSonic Endovascular System with thrombolytic

INTERVENTIONS:
Device: EkoSonic Endovascular System with thrombolytic — The device uses ultrasonic waves in combination with clot-dissolving thrombolytic drug to effectively dissolve clots.
  Other Names: Acoustic Pulse Thrombolysis; EKOS

SUMMARY:
This registry is designed to understand acoustic pulse thrombolysis (APT) treatment regimens used as standard of care globally for pulmonary embolism. The registry will include individuals who have already received the APT treatment and those that will undergo APT treatment.

DETAILED DESCRIPTION:
For the prospective arm of the registry, a physician will have selected the APT procedure for the treatment of pulmonary embolism. The APT treatment and follow-up assessments are per clinical judgement and institutional standard of care which may vary at each clinical site.

For the retrospective arm of the registry, the investigators will gather data from consecutive cases of individuals who received the APT treatment for pulmonary embolism. Specific baseline, treatment, and long-term health information is collected and de-identified.

ELIGIBILITY:
Retrospective Inclusion Criteria:

* Treated with APT procedure between January 1, 2014 and one year prior to site activation
* RV/LV ≥ 1.0 from diagnostic computed tomographic angiography (CTA) or echocardiogram
* PE symptom duration ≤ 14 days
* Troponin elevation

Retrospective Exclusion Criteria:

* Enrollment into the OPTALYSE PE study

Prospective Inclusion Criteria:

* Male or female ≥ 18 years of age and ≤ 80 years of age
* RV/LV ≥ 1.0 from diagnostic computed tomographic angiography (CTA) or echocardiogram
* PE symptom duration ≤ 14 days
* Troponin elevation
* Signed informed consent obtained from participant or legally authorized representative
* Investigator has selected the EKOS device to treat participant with massive or submassive pulmonary embolism

Prospective Exclusion Criteria:

* High-risk for catastrophic bleeding
* Life expectancy < one year

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals with intermediate-high and high risk pulmonary embolism who are selected to receive treatment using the EKOS device and thrombolytic.
Sampling Method: Non-Probability Sample
Enrollment: 1480 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Keith Sterling, MD, Principal Investigator — Inova Alexandria Hospital
Locations (80):
- United States (65):
  - Healthfinity, PLLC Advanced Cardiac & Vascular Clinic, Glendale, Arizona
  - Cedars - Sinai, Los Angeles, California
  - Radiology Imaging Associates, Englewood, Colorado
  - Bradenton Cardiology Center, Bradenton, Florida
  - Delray Medical Center, Delray Beach, Florida
  - St. Vincent's Healthcare, Jacksonville, Florida
  - University of Florida, Jacksonville, Florida
  - Memorial Hospital, Jacksonville, Florida
  - University of Miami, Miami, Florida
  - Florida Hospital, Orlando, Florida
  - Orlando Health, Inc., Orlando, Florida
  - Tallahassee Research Institute, Inc, Tallahassee, Florida
  - AdventHealth Tampa Pepin Heart Institute, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - Augusta University, Augusta, Georgia
  - WellStar Medical Group, Marietta, Georgia
  - Northwestern University, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - St. Mary Medical Center, Hobart, Indiana
  - St. Vincent Hospital, Indianapolis, Indiana
  - St. Elizabeth Healthcare, Crestview Hills, Kentucky
  - University of Kentucky, Lexington, Kentucky
  - Jewish Hospital, Louisville, Kentucky
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham & Women's Hospital, Boston, Massachusetts
  - St. Vincent Hospital/Reliant Medical Group, Worcester, Massachusetts
  - University of Michigan Health System, Ann Arbor, Michigan
  - Ascension St. John Hospital, Detroit, Michigan
  - Spectrum Health, Grand Rapids, Michigan
  - Metro Health - University of Michigan Health, Wyoming, Michigan
  - Cardiology Associates of Northern Mississippi, Oxford, Mississippi
  - Saint Louis University Hospital, St Louis, Missouri
  - Dartmouth - Hitchcock Medical Center, Lebanon, New Hampshire
  - Cooper University Healthcare, Camden, New Jersey
  - University of Buffalo, Buffalo, New York
  - Duke University Medical Center, Durham, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - Summa Health, Akron, Ohio
  - Mercy Health Cincinnati, Cincinnati, Ohio
  - University of Cincinnati, Cincinnati, Ohio
  - TriHealth Good Samaritan Bethesda North, Cincinnati, Ohio
  - Ohio State University, Columbus, Ohio
  - Mount Caramel East Hospital, Columbus, Ohio
  - University of Toledo, Toledo, Ohio
  - Genesis Healthcare System, Zanesville, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - St. Luke's University Health Network, Bethlehem, Pennsylvania
  - St. Vincent Hospital, Allegheny Health Network, Erie, Pennsylvania
  - Temple University Hospital, Department of Thoracic Medicine & Surgery, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - UPMC Hamot, Pittsburgh, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - Lexington Cardiology, West Columbia, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Hendrick Medical Center, Abilene, Texas
  - The Heart Hospital Baylor Plano, Plano, Texas
  - Houston Methodist Sugarland, Sugar Land, Texas
  - Inova Alexandria Hospital, Alexandria, Virginia
  - Sentara Vascular Specialists, Norfolk, Virginia
  - Providence Regional Medical Center, Everett, Washington
  - Inland Imaging, Spokane, Washington
  - CAMC, Charleston, West Virginia
  - West Virginia University Heart & Vascular Institute, Morgantown, West Virginia
  - Aurora Cardiovascular Services, Milwaukee, Wisconsin
- Medical University of Vienna, Vienna, Austria
- France (2):
  - CHRU jean Minjoz, Pôle cœur-Poumons, Besançon
  - Hôpital Nord, APHM, Marseille
- Germany (2):
  - Johannes Gutenberg Univeristy Mainz, Mainz
  - Technical University Munchen, München
- University Medical Center Uterecht, Utrecht, Netherlands
- Switzerland (2):
  - Swiss Cardiovascular Center, Bern
  - University Hospital Zurich, Zurich
- Acibadem University School of Medicine, Istanbul, Turkey (Türkiye)
- United Kingdom (6):
  - Royal Devon and Exeter Hospital, Exeter
  - Medway NHS Foundation Trust, Gillingham
  - Oxford University Hospitals, Headington
  - Royal Free, London
  - Guy's & St Thomas' NHS Foundation Trust, London
  - St. Mary's Hospital, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sterling KM, Goldhaber SZ, Sharp ASP, Kucher N, Jones N, Maholic R, Meneveau N, Zlotnick D, Sayfo S, Konstantinides SV, Piazza G. Prospective Multicenter International Registry of Ultrasound-Facilitated Catheter-Directed Thrombolysis in Intermediate-High and High-Risk Pulmonary Embolism (KNOCOUT PE). Circ Cardiovasc Interv. 2024 Mar;17(3):e013448. doi: 10.1161/CIRCINTERVENTIONS.123.013448. Epub 2024 Jan 24. PMID 38264938

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Retrospective | Prospective
Started | 991 | 489
Completed | 941 | 251
Not Completed | 50 | 238

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Retrospective | Prospective | Total
Number analyzed (Participants) | 991 | 489 | 1480
Age, Continuous [Median (Full Range); unit: years] | 62.0 [14 to 93] | 63.0 [20 to 81] | 63.0 [20 to 81]
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 486 | 259 | 745
  Female | 504 | 230 | 734
  No Answer | 1 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 652 | 296 | 948
  African American | 192 | 77 | 269
  Other | 13 | 9 | 22
  Unknown or Missing | 134 | 117 | 251
Baseline Medical History [Count of Participants; unit: Participants]
  Active Cancer | 79 | 20 | 99
  BMI ≥30.0 kg/m² | 642 | 319 | 961
  Family History of Venous Thromboembolism | 109 | 71 | 180
  History of Cancer in Remission | 116 | 60 | 176
  Congestive Heart Failure | 54 | 13 | 67

OUTCOME MEASURES:

1. Primary Outcome: Change in RV/LV Ratio on Echocardiogram (Matched Pairs as Available)
Description: Difference (percent change) in the measurement of the right ventricular to left ventricular diameters (RV/LV) ratio as measured on baseline echocardiogram to post-procedure echocardiogram (24-48 hours post initiation of therapy).
Time Frame: Baseline to post-procedure (end of procedure through hospital discharge up to 14 days)
Population: Subjects with matched pairs (pre-procedure echocardiogram and post-procedure echocardiogram through discharge from index hospitalization) have been reported.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Retrospective | Prospective
Number analyzed (Participants) | 276 | 176
Percent change | -22.6 (20.8) | -22.6 (19.9)

2. Primary Outcome: Frequency and Safety Outcomes of Subjects Requiring Interventions of Adjunctive Therapies Post-procedure During Hospitalization.
Description: Measured by number of subjects requiring interventions of adjunctive therapies received during post procedure hospitalization through hospital discharge up to 14 days.
Time Frame: Post-procedure hospitalization through hospital discharge up to 14 days
Measure: Count of Participants; unit: Participants
Arm/Group | Retrospective | Prospective
Number analyzed (Participants) | 991 | 489
Participants
  Continuation of procedure beyond planned time/dose | 7 | 1
  Surgical pulmonary embolectomy | 0 | 1
  Catheter-assisted embolectomy including thrombus fragmentation or aspiration | 5 | 2
  Peripherally administered systemic fibrinolytic therapy | 4 | 0
  Other therapy/procedure | 40 | 3

3. Primary Outcome: Number of Patients Who Underwent Interventional Therapies Prior to the APT Procedure and Experienced a Non- or Partial- Response.
Description: Measured by number of patients who underwent interventional therapies prior to the APT procedure and experienced a non or partial response.
Time Frame: From date of enrollment up to or until the placement of the Ekos device, on average 48 hours.
Measure: Count of Participants; unit: Participants
Arm/Group | Retrospective | Prospective
Number analyzed (Participants) | 991 | 489
Participants
  Peripherally administered systemic fibrinolytic therapy | 9 | 1
  Surgical pulmonary embolectomy | 5 | 0
  Catheter-assisted embolectomy including fragmentation or aspiration | 19 | 0
  Other | 11 | 3

4. Primary Outcome: Number of Patients Experiencing a SAEs Related to EKOS Device and/or Procedure During First 12 Months Post-APT Procedure.
Description: Number of subjects experiencing a SAE related to EKOS device and/or procedure from time of procedure through the first 12 months post-APT procedure, measured by frequency and severity of events.
Time Frame: From time of APT procedure through 12 months post-procedure.
Measure: Count of Participants; unit: Participants
Arm/Group | Retrospective | Prospective
Number analyzed (Participants) | 991 | 489
Participants
  SAEs related to EKOS device and/or procedure - Severe | 9 | 5
  SAEs related to EKOS device and/or procedure - Moderate | 6 | 1
  SAEs related to EKOS device and/or procedure - Mild | 1 | 0

5. Primary Outcome: All-cause Mortality During First 12 Months Post-procedure.
Description: Number of all-cause mortality that occurred from the start of procedure through 12 months post-procedure.
Time Frame: Start of procedure through 12 months post-procedure.
Population: Retrospective data to be updated.
Measure: Count of Participants; unit: Participants
Arm/Group | Retrospective | Prospective
Number analyzed (Participants) | 991 | 489
Participants | 50 | 15

6. Primary Outcome: Healthcare Utilization
Description: Summary of healthcare utilization from date of enrollment through discharge.
Time Frame: Measured as time from ICU admission to ICU discharge in hours (from date of enrollment through 12 months post-procedure).
Measure: Median (Inter-Quartile Range); unit: Hours
Arm/Group | Retrospective | Prospective
Number analyzed (Participants) | 991 | 483
Hours | 44.2 [27.3 to 64.6] | 41.2 [25.8 to 54.3]

7. Primary Outcome: Change in Quality of Life (QOL) as Measured by the Pulmonary Embolism Quality of Life (PEmb-QOL) at the 3 Month and 12 Month Post-hospitalization Follow-up Visits
Description: Reported as percent change in the PEmb-QOL questionnaire score from baseline timepoint to 3 months and 12 months. The PEmb-QOL measures patient's quality of life following pulmonary embolism on a scale of 1 through 5, with lower scores indicating a better outcome.
Time Frame: Measured as percent change in time from baseline assessment at discharge to 3 month and 12 month follow up.
Population: QOL date were not collected in the retrospective cohort. These questionnaires were only collected prospectively.
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Retrospective | Prospective
Number analyzed (Participants) | 0 | 243
percentage change
  PEmb-QOL Mean Change at 3 Months |  | -22.52 (24.12)
  PEmb-QOL Mean Change at 12 Months |  | -23.74 (24.14)

8. Primary Outcome: Change in Quality of Life (QOL) as Measured by the EQ-5D-5L VAS, Utility and Misery Scores at the 3-month and 12-month Post-hospitalization Follow-up Visits.
Description: Reported as change in the VAS, Utility and Misery questionnaire scores from baseline timepoint and/or study visit to 3 months and 12 months.
  The VAS (Visual Analogue Scale) is a one question, unidimensional measure of pain intensity where a subject is asked to rate his pain on a scale of 100 through 1, with 100 indicating the best health imaginable through 1 indicating the worst health imaginable. Higher scores indicate a better outcome.
  The EQ-5D is a series of questions that measures Quality of Life on a scale of 0 through 5. 0 indicates no problems in daily activities and 5 indicates inability to perform daily activities. The total score is added up and compared to the total scale from 0 to 25, with 0 indicating no problems in daily activities and 25 indicating inability to perform daily activities. A lower score indicates a better outcome.
Time Frame: Reported results include change from baseline to 3 months and 12 months post-procedure for prospective patients.
Population: Data for the retrospective cohort were not captured as Quality of Life questionnaires were not Standard of Care at most institutions.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Retrospective | Prospective
Number analyzed (Participants) | 0 | 483
units on a scale
  Change in VAS at 3 Months: number analyzed (Participants) | 0 | 242
  Change in VAS at 3 Months |  | 12.4 (24.36)
  Change in VAS at 12 Months: number analyzed (Participants) | 0 | 152
  Change in VAS at 12 Months |  | 11.1 (21.7)
  Change in Utility Score at 3 Months: number analyzed (Participants) | 0 | 243
  Change in Utility Score at 3 Months |  | 0.20 (0.35)
  Change in Utility Score at 12 Months: number analyzed (Participants) | 0 | 152
  Change in Utility Score at 12 Months |  | 0.19 (0.31)
  Change in Misery Score at 3 Months: number analyzed (Participants) | 0 | 243
  Change in Misery Score at 3 Months |  | -2.8 (4.8)
  Change in Misery Score at 12 Months: number analyzed (Participants) | 0 | 152
  Change in Misery Score at 12 Months |  | -2.7 (4.3)

9. Primary Outcome: Number of Patients Needing an IVC Filter Placement
Description: Measured by number patients with an occurrence of needing an IVC filter placement.
Time Frame: From date of procedure through 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Retrospective | Prospective
Number analyzed (Participants) | 991 | 483
Participants | 50 | 20

10. Primary Outcome: Number of Patients Experiencing Adverse Events Classified as Major Bleeding Events During First 12 Months Post-Procedure by Frequency and Severity
Description: Measured by number of patients experiencing adverse events related to major bleeding events from time of procedure through the first 12 months post-procedure by frequency and severity (mild, moderate, severe).
Time Frame: From post-procedure through 12-months post-procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Retrospective | Prospective
Number analyzed (Participants) | 991 | 489
Participants
  Major Bleeds within 365 days - Mild | 10 | 3
  Major Bleeds within 365 days - Moderate | 33 | 8
  Major Bleeds within 365 days - Severe | 18 | 3

11. Primary Outcome: Number of Patients Experiencing VTE (Venus Thromboembolytic Events) During First 12 Months Post-Procedure by Frequency and Severity.
Description: Number of patients experiencing events related to VTE from time of procedure through the first 12 months post-procedure by frequency and severity.
Time Frame: From post-procedure through 12-months post-procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Retrospective | Prospective
Number analyzed (Participants) | 991 | 489
Participants
  VTEs within 365 Days - Mild | 33 | 31
  VTEs within 365 Days - Moderate | 15 | 11
  VTEs within 365 Days - Severe | 15 | 5

12. Primary Outcome: Diagnosis of Pulmonary Hypertension Diagnosis
Description: New onset pulmonary hypertension defined as mean pulmonary artery pressure greater than 25 mm Hg by echocardiogram that persists at least 3 months after PE.
Time Frame: Analyzed 12 months post-procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Retrospective | Prospective
Number analyzed (Participants) | 991 | 489
Participants | 0 | 1

ADVERSE EVENTS:
Time Frame: Adverse Events were collected on or after the date of the procedure through 12 months. Data presented are for prospective and retrospective patients through the 12 month follow up visit.
Description: Only TEAEs (Treatment Emergent Adverse Event), defined as AEs starting on or after the date of intervention are included in this table. Patients are counted at most once for each preferred MedDRA term. Some patients were not followed for the full 12 months due to retrospective data collection and prospective data collection ending prior to the last patient reaching 12 months.
Arm/Group | Retrospective | Prospective
All-Cause Mortality (participants affected / at risk) | 50/991 | 15/489
Serious Adverse Events (participants affected / at risk) | 100/991 | 39/489
Other Adverse Events (participants affected / at risk) | 63/991 | 40/489
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Retrospective (N=991) | Prospective (N=489)
Anaemia (Blood and lymphatic system disorders) | 4 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Atrial Fibrillation (Cardiac disorders) | 0 | 0
Atroventricular block, complete (Cardiac disorders) | 1 | 0
Bradycardia (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 10 | 0
Cardiac tamponade (Cardiac disorders) | 0 | 1
Cardiogenic shock (Cardiac disorders) | 1 | 0
Dyspnoea (Cardiac disorders) | 0 | 1
Endocarditis, bacterial (Cardiac disorders) | 1 | 0
Pulseless electrical activity (Cardiac disorders) | 3 | 0
Reperfusion arrhythmia (Cardiac disorders) | 1 | 0
Right ventricular failure (Cardiac disorders) | 1 | 0
Diverticulum (Gastrointestinal disorders) | 1 | 0
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 1
Death (General disorders) | 3 | 5
Multiple organ dysfunction syndrome (General disorders) | 1 | 2
Pneumonia (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 2 | 0
Soft tissue infection (Infections and infestations) | 0 | 1
Gun shot wound (Injury, poisoning and procedural complications) | 0 | 1
Traumatic haematoma (Injury, poisoning and procedural complications) | 1 | 0
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Astrocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon cancer, metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung cancer, metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastatic renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neoplasm, malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Neuroendocrine tumor (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Subdural haematoma (Nervous system disorders) | 1 | 0
Delirium (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cardio-respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Chronic pulmonary obstructive disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Abdominal wall haemorrhage (Vascular disorders) | 1 | 0
Acute myocardial infarction (Vascular disorders) | 1 | 1
Cardiogenic shock (Vascular disorders) | 2 | 0
Cerebellar haemorrhage (Vascular disorders) | 1 | 0
Cerebral haemorrhage (Vascular disorders) | 2 | 0
Cerebral infarction (Vascular disorders) | 1 | 0
Cerebrovascular accident (Vascular disorders) | 1 | 0
Compartment syndrome (Vascular disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 5 | 1
Disseminated intravascular coagulation (Vascular disorders) | 2 | 0
Embolism, venous (Vascular disorders) | 1 | 1
Gastrointestinal haemorrhage (Vascular disorders) | 5 | 1
Haematochezia (Vascular disorders) | 1 | 0
Haematoma (Vascular disorders) | 7 | 0
Haematuria (Vascular disorders) | 1 | 1
Haemoptysis (Vascular disorders) | 0 | 1
Haemorrhage (Vascular disorders) | 1 | 0
Haemorrhage, intracranial (Vascular disorders) | 3 | 0
Heparin-induced thrombocytopenia (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0
Hypoxic-ischaemic encephalopathy (Vascular disorders) | 1 | 0
Internal haemorrhage (Vascular disorders) | 1 | 0
Lacunar infarction (Vascular disorders) | 1 | 0
Lower gastrointestinal haemorrhage (Vascular disorders) | 1 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 1 | 0
Post procedural haematoma (Vascular disorders) | 1 | 0
Post procedural haemorrhage (Vascular disorders) | 2 | 0
Pulmonary embolism (Vascular disorders) | 12 | 7
Pulmonary hypertension (Vascular disorders) | 1 | 2
Retroperitoneal haematoma (Vascular disorders) | 1 | 0
Retroperitoneal haemorrhage (Vascular disorders) | 0 | 1
Shock, hemorrhagic (Vascular disorders) | 1 | 0
Subdural haematoma (Vascular disorders) | 1 | 1
Transient ischaemic attack (Vascular disorders) | 1 | 0
Vaginal hemorrhage (Vascular disorders) | 1 | 1
Vascular access site haematoma (Vascular disorders) | 0 | 1
Vascular pseudoaneurysm (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Retrospective (N=991) | Prospective (N=489)
Deep Vein Thrombosis (Vascular disorders) | 39 | 34
Haematoma (Vascular disorders) | 24 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-10-19): https://cdn.clinicaltrials.gov/large-docs/24/NCT03426124/Prot_000.pdf
  • Statistical Analysis Plan (2019-03-01): https://cdn.clinicaltrials.gov/large-docs/24/NCT03426124/SAP_001.pdf